CLINICAL TRIAL: NCT03266302
Title: Revealing Mechanisms and Investigating Efficacy of Hemoadsorption for Prevention of Vasodilatory Shock in Cardiac Surgery Patients With Infective Endocarditis - a Multicentric Randomized Controlled Group Sequential Trial
Brief Title: Hemoadsorption for Prevention of Vasodilatory Shock in Cardiac Surgery Patients With Infective Endocarditis
Acronym: REMOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: CytoSorbents, Inc (Industry); Thermo Fisher Scientific, Inc (Industry); Fraunhofer Institute for Interfacial Engineering and Biotechnology (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: ZKSJ0108
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2020-03

CONDITIONS: Infective Endocarditis
Keywords: vasodilatory shock; hemoadsorption; cardiac surgery; cytokines
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Intervention Model Description: two-arm randomized-controlled group sequential (Pocock) design for assessing superiority and safety
Who Masked: Participant
Masking Description: Participant will not be informed about group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Use of hemoadsorber for removal of cytokines. Participants undergoing cardiac surgery due to infective endocarditis will be treated using a hemoadsorption device (CytoSorb) within the cardiopulmonary Bypass circuit (=Intervention)
  Interventions: Device: hemoadsorber for removal of cytokines
- Control group (No Intervention): Participants undergoing cardiac surgery due to infective endocarditis will be treated according to Standard of care (no hemoadsorption advice installed in the CPB circuit)

INTERVENTIONS:
Device: hemoadsorber for removal of cytokines — Use of the hemoadsorber during cardiac surgery with CPB. Hemoadsorber is integrated into the CPB circuit according to manufacturer's recommendation.
  Other Names: CytoSorb(R)
  Arms: Interventional group

SUMMARY:
Infective endocarditis (IE) is associated with high hospital mortality for various reasons; one of them is circulatory failure in patients who undergo cardiac surgery for IE. One discussed reason underlying circulatory failure during surgery is the release of vasodilatatory mediators and cytokines. This study examines the efficacy and safety of a hemoadsorption filter which is approved for the reduction of the concentration of cytokines in the bloodstream.

DETAILED DESCRIPTION:
The investigators assume a common standard deviation of 3.8 points and that a 1.4-point lower SOFA score in the Intervention Group is of clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* patients with infective endocarditis (according to DUKE criteria) undergoing cardiac surgery
* informed consent
* age ≥18 years

Exclusion Criteria:

* EuroScoreII ≤ 3
* current participation in another interventional Trial
* pregnancy
* current immunosuppressive or immunomodulatory therapy (with dosing of glucocorticoids over Cushing threshold)
* previous participation in the REMOVE study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
SOFA Score | 24 hours before until day 9 post-surgery
  The investigators will test if mean SOFA scores are different for the experimental and control group.

SECONDARY OUTCOMES:
Overall mortality rate | until day 30 post surgery
  Overall mortality rate until day 30 post-surgery
Changes in cytokine and cfDNA levels | 24 hours before, during cardiac surgery and 24 hours after surgery
  changes in cytokine and cfDNA levels will be measured at different time points before, during and after surgery in both groups; only for the first 2x25 patients
SOFA subscores | 24 hours before surgery until day 9 post-surgery
  single SOFA subscores will be analyzed
Days on ventilator, vasopressor and renal replacement therapy | until day 30 post-surgery
  Total days on ventilator, vasopressor and renal replacement therapy within 30 days post-surgery will be assessed
incidence of stroke | until day 30 post-surgery
  incidence of stroke within 30 days post-surgery will be assessed
length of ICU and in-hospital stay | until day 30 post-surgery
  total length of ICU and in-hospital stay until day 30 post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Diab, Dr., Study Director — Jena University Hospital, Department of Cardiac and Thoracic Surgery
Locations (14):
- Germany (14):
  - University Heart Center Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - University Heart Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Hospital Ulm, Clinics of Heart-, Thoracic and Cardiovascular Surgery, Ulm, Baden-Wurttemberg
  - University Hospital Cologne, Clinic and Policlinics for Heart and Thoracic Surgery, Cologne, North Rhine-Westphalia
  - University Hospital Essen, Clinic of Thoracic and Cardiovascular Surgery, Essen, North Rhine-Westphalia
  - Jena University Hospital, Dept. of Cardiac and Thoracic Surgery, Jena, Thuringia
  - Herz- und Diabeteszentrum NRW, Klinik für Thorax- und Kardiovaskularchirurgie, Bad Oeynhausen
  - Herzzentrum Brandenburg, Immanuel Klinikum Bernau, Bernau bei Berlin
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil gGmbH, Klinik für Herz- und Thoraxchirurgie, Bochum
  - Universitätsklinikum Bonn, Klinik und Poliklinik für Herzchirurgie, Bonn
  - Herzzentrum Dresden GmbH, Universitätsklinik an der TU Dresden, Klinik für Herzchirurgie, Dresden
  - Universitätsklinikum Düsseldorf, Klinik für Kardiovaskuläre Chirurgie, Düsseldorf
  - Mitteldeutsches Herzzentrum, Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Herzchirurgie, Halle
  - Herzzentrum Leipzig, Universitätsklinik für Herzchirurgie, Leipzig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernardi MH, Rinoesl H, Dragosits K, Ristl R, Hoffelner F, Opfermann P, Lamm C, Preissing F, Wiedemann D, Hiesmayr MJ, Spittler A. Effect of hemoadsorption during cardiopulmonary bypass surgery - a blinded, randomized, controlled pilot study using a novel adsorbent. Crit Care. 2016 Apr 9;20:96. doi: 10.1186/s13054-016-1270-0. PMID 27059056
- [Background] Brunkhorst FM, Oppert M, Marx G, Bloos F, Ludewig K, Putensen C, Nierhaus A, Jaschinski U, Meier-Hellmann A, Weyland A, Grundling M, Moerer O, Riessen R, Seibel A, Ragaller M, Buchler MW, John S, Bach F, Spies C, Reill L, Fritz H, Kiehntopf M, Kuhnt E, Bogatsch H, Engel C, Loeffler M, Kollef MH, Reinhart K, Welte T; German Study Group Competence Network Sepsis (SepNet). Effect of empirical treatment with moxifloxacin and meropenem vs meropenem on sepsis-related organ dysfunction in patients with severe sepsis: a randomized trial. JAMA. 2012 Jun 13;307(22):2390-9. doi: 10.1001/jama.2012.5833. PMID 22692171
- [Background] Bustamante J, Arevalo A, Tamayo E, Sarria C, Aguilar-Blanco EM, Heredia M, Almansa R, Rico L, Iglesias V, Bermejo-Martin JF. Cytokine profiles linked to fatal outcome in infective prosthetic valve endocarditis. APMIS. 2014 Jun;122(6):526-9. doi: 10.1111/apm.12189. Epub 2013 Sep 30. PMID 24106887
- [Background] Boyle EM Jr, Pohlman TH, Johnson MC, Verrier ED. Endothelial cell injury in cardiovascular surgery: the systemic inflammatory response. Ann Thorac Surg. 1997 Jan;63(1):277-84. doi: 10.1016/s0003-4975(96)01061-2. PMID 8993292
- [Background] Hotchkiss RS, Karl IE. The pathophysiology and treatment of sepsis. N Engl J Med. 2003 Jan 9;348(2):138-50. doi: 10.1056/NEJMra021333. No abstract available. PMID 12519925
- [Background] Minne L, Abu-Hanna A, de Jonge E. Evaluation of SOFA-based models for predicting mortality in the ICU: A systematic review. Crit Care. 2008;12(6):R161. doi: 10.1186/cc7160. Epub 2008 Dec 17. PMID 19091120
- [Background] Prendergast BD, Tornos P. Surgery for infective endocarditis: who and when? Circulation. 2010 Mar 9;121(9):1141-52. doi: 10.1161/CIRCULATIONAHA.108.773598. No abstract available. PMID 20212293
- [Result] Diab M, Lehmann T, Bothe W, Akhyari P, Platzer S, Wendt D, Deppe AC, Strauch J, Hagel S, Gunther A, Faerber G, Sponholz C, Franz M, Scherag A, Velichkov I, Silaschi M, Fassl J, Hofmann B, Lehmann S, Schramm R, Fritz G, Szabo G, Wahlers T, Matschke K, Lichtenberg A, Pletz MW, Gummert JF, Beyersdorf F, Hagl C, Borger MA, Bauer M, Brunkhorst FM, Doenst T; REMOVE Trial Investigators*. Cytokine Hemoadsorption During Cardiac Surgery Versus Standard Surgical Care for Infective Endocarditis (REMOVE): Results From a Multicenter Randomized Controlled Trial. Circulation. 2022 Mar 29;145(13):959-968. doi: 10.1161/CIRCULATIONAHA.121.056940. Epub 2022 Feb 25. PMID 35213213
- [Derived] Diab M, Platzer S, Guenther A, Sponholz C, Scherag A, Lehmann T, Velichkov I, Hagel S, Bauer M, Brunkhorst FM, Doenst T. Assessing efficacy of CytoSorb haemoadsorber for prevention of organ dysfunction in cardiac surgery patients with infective endocarditis: REMOVE-protocol for randomised controlled trial. BMJ Open. 2020 Mar 30;10(3):e031912. doi: 10.1136/bmjopen-2019-031912. PMID 32234739